CLINICAL TRIAL: NCT03989232
Title: Efficacy and Safety of Semaglutide 2.0 mg s.c. Once-weekly Compared to Semaglutide 1.0 mg s.c. Once-weekly in Subjects With Type 2 Diabetes
Brief Title: A Research Study to Compare Two Doses of Semaglutide Taken Once Weekly in People With Type 2 Diabetes
Acronym: SUSTAIN FORTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-4506; U1111-1224-5162 (Other: World Health Organization (WHO)); 2018-004529-96 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide 2.0 mg (Experimental): All participants will receive one injection per week during a 12-week dose escalation period, until the target dose for semaglutide 2.0 mg is reached. From week 13 to week 40, semaglutide will be given in two weekly injections of 1.0 mg each.
  Interventions: Drug: Semaglutide
- Semaglutide 1.0 mg (Active Comparator): All participants will receive one injection per week during a 12-week dose escalation period. From week 13 to week 40, the 1.0 mg group will receive an additional injection of semaglutide placebo in order to maintain the blinding.
  Interventions: Drug: Semaglutide; Drug: Placebo (semaglutide)

INTERVENTIONS:
Drug: Semaglutide — Semaglutide injected subcutaneously (s.c., under the skin) once-weekly. Participants will keep taking their pre-study diabetes tablets throughout the study.
Drug: Placebo (semaglutide) — Semaglutide placebo injected once-weekly from week 13 to week 40.
  Arms: Semaglutide 1.0 mg

SUMMARY:
This study compares the effect of two doses of semaglutide (1.0 mg and 2.0 mg) in people with type 2 diabetes (T2D). People taking part in the study will take the medicine together with their current diabetes medicine (sulphonylurea and/or metformin). Participants will get a dose of either 1.0 mg or 2.0 mg semaglutide once a week - which dose is decided by chance. Participants will inject semaglutide under the skin once a week. The study will last for about 49 weeks. Participants will have 9 clinic visits and 2 phone calls with the study doctor. At the visits participants will have blood taken and eye tests done. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period. Female participants who can get pregnant will be checked 11 times for pregnancy via urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age equal to or above18 years at the time of signing informed consent
* Diagnosed with T2D at least 180 days prior to the day of screening
* HbA1c of 8-10% (64-86 mmol/mol) (both inclusive)
* Stable daily dose(s) for 90 days prior to the day of screening of:
* Any metformin formulations (equal to or above1500 mg or maximum tolerated or effective dose) alone or in combination with sulfonylureas (SU) (equal to or above half of the maximum approved dose according to local label or maximum tolerated or effective dose)

Exclusion Criteria:

* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes
* Renal impairment measured as estimated glomerular filtration rate (eGFR) value of <30 mL/min/1.73 m^2 according to the Chronic Kidney Disease Epidemiology Collaboration (CKDEPI) creatinine equation as defined by KDIGO 2012 classification
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 961 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (108):
- United States (58):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Chandler, Arizona
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Buena Park, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, West Hills, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Coral Gables, Florida
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Adairsville, Georgia
  - Novo Nordisk Investigational Site, Alpharetta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Carlinville, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Lake Charles, Louisiana
  - Novo Nordisk Investigational Site, Sterling Heights, Michigan
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Trenton, New Jersey
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Salisbury, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Corvallis, Oregon
  - Novo Nordisk Investigational Site, Gaffney, South Carolina
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Humble, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Shavano Park, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Walla Walla, Washington
  - Novo Nordisk Investigational Site, Wenatchee, Washington
- Bulgaria (6):
  - Novo Nordisk Investigational Site, Kozloduy
  - Novo Nordisk Investigational Site, Montana
  - Novo Nordisk Investigational Site, Petrich
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Stara Zagora
  - Novo Nordisk Investigational Site, Yambol
- Canada (7):
  - Novo Nordisk Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Markham, Ontario
  - Novo Nordisk Investigational Site, Stoney Creek, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
- Czechia (3):
  - Novo Nordisk Investigational Site, České Budějovice
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Vlašim
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (6):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Kaposvár
  - Novo Nordisk Investigational Site, Komárom
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Szekszárd
- Novo Nordisk Investigational Site, Tokyo, Japan
- Poland (8):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Gorzów Wielkopolski
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Novo Nordisk Investigational Site, Manatí, Puerto Rico
- Slovakia (11):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Hnúšťa
  - Novo Nordisk Investigational Site, Kežmarok
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Krupina
  - Novo Nordisk Investigational Site, Levice
  - Novo Nordisk Investigational Site, Nové Zámky
  - Novo Nordisk Investigational Site, Pezinok
  - Novo Nordisk Investigational Site, Poprad
  - Novo Nordisk Investigational Site, Považská Bystrica
  - Novo Nordisk Investigational Site, Púchov
- Ukraine (5):
  - Novo Nordisk Investigational Site, Dnipro
  - Novo Nordisk Investigational Site, Mykolaiv
  - Novo Nordisk Investigational Site, Ternopil
  - Novo Nordisk Investigational Site, Vinnytsia
  - Novo Nordisk Investigational Site, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Frias JP, Auerbach P, Bajaj HS, Fukushima Y, Lingvay I, Macura S, Sondergaard AL, Tankova TI, Tentolouris N, Buse JB. Efficacy and safety of once-weekly semaglutide 2.0 mg versus 1.0 mg in patients with type 2 diabetes (SUSTAIN FORTE): a double-blind, randomised, phase 3B trial. Lancet Diabetes Endocrinol. 2021 Sep;9(9):563-574. doi: 10.1016/S2213-8587(21)00174-1. Epub 2021 Jul 21. PMID 34293304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 125 sites in Bulgaria (9), Canada (8), Czech Republic (4), Greece (6), Hungary (12), Japan (2), Poland (10), Slovakia (11), Ukraine (5) and the United States (58). In addition to these sites, 4 sites in the US screened but did not randomize participants, and 3 sites were approved by the IRB/IEC but did not screen or assign any participants to treatment.
Pre-assignment Details: Participants with type 2 diabetes (T2D) treated with stable doses of metformin only, or metformin in combination with sulfonylurea (SU), in need of the treatment intensification were randomized 1:1 to once-weekly treatment with semaglutide 2.0 milligrams (mg) or once-weekly treatment with semaglutide 1.0 mg.
Groups:
- Semaglutide 1.0 mg: Participants received subcutaneous (s.c.) injection of semaglutide once-weekly for 40 weeks in a fixed-dose escalation regimen, with dose doubling every 4 weeks until the target dose of 1.0 mg was reached: 0.25 mg during 0-4 weeks followed by 0.5 mg during 4-8 weeks followed by 1.0 mg during 8-12 weeks and then 1.0 mg semaglutide along with s.c. injection of placebo matched to semaglutide 1.0 mg during 12-40 weeks.
- Semaglutide 2.0 mg: Participants received s.c. injection of semaglutide once-weekly for 40 weeks in a fixed-dose escalation regimen, with dose doubling every 4 weeks until the target maintenance dose of 2.0 mg was reached: 0.25 mg during 0-4 weeks followed by 0.5 mg during 4-8 weeks followed by 1.0 mg during 8-12 weeks and then 2.0 mg during 12-40 weeks.
Period: Overall Study
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Started | 481 | 480
Exposed | 480 | 479
Safety Analysis Set (SAS) | 480 | 479
Full Analysis Set (FAS) | 481 | 480
Completed | 471 | 462
Not Completed | 10 | 18
Not completed — Lost to Follow-up | 3 | 10
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg | Total
Number analyzed (Participants) | 481 | 480 | 961
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (9.9) | 57.9 (10.0) | 58.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 201 | 398
  Male | 284 | 279 | 563
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 52 | 111
  Not Hispanic or Latino | 422 | 428 | 850
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska native | 1 | 0 | 1
    Asian | 36 | 33 | 69
    Black or African American | 17 | 26 | 43
    Native Hawaiian or Other Pacific | 0 | 0 | 0
    White | 427 | 420 | 847
    Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change from baseline (week 0) to week 40 in glycosylated haemoglobin (HbA1c) was evaluated.
  Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first; and 'In-trial' observation period which started at the date of randomisation and ended at the first of the following dates, both inclusive: end-of-treatment visit (week 40), death, participant withdrew informed consent, last contact for participant lost to follow-up.
Time Frame: Week 0, week 40
Population: The FAS included all randomized participants. Number analyzed=number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 481 | 480
Percentage change
  On-treatment without rescue medication: number analyzed (Participants) | 422 | 423
  On-treatment without rescue medication | -2.0 (1.0) | -2.2 (1.0)
  In-trial: number analyzed (Participants) | 466 | 456
  In-trial | -1.9 (1.0) | -2.2 (1.1)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Semaglutide 2.0 mg; On-treatment without rescue medication observation period: Imputation of missing data was handled by multiple imputation (MI) assuming that missing data were missed at random (MAR). The imputation was performed separately within each treatment group defined by randomised treatment; Test type: Superiority; p = 0.0003, ANCOVA; Treatment difference = -0.23, 95% CI 2-sided [-0.36 to -0.11]
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Semaglutide 2.0 mg; In-trial observation period: Imputation of missing data was handled by MI assuming that missing data were missed at random. The imputation was performed by imputing missing week 40 data separately within groups defined by randomised treatment and treatment status at week 40; Test type: Superiority; p = 0.0098, ANCOVA; Treatment difference = -0.18, 95% CI 2-sided [-0.31 to -0.04]

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) to week 40 in body weight was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first; and 'In-trial' observation period which started at the date of randomisation and ended at the first of the following dates, both inclusive: end-of-treatment visit (week 40), death, participant withdrew informed consent, last contact for participant lost to follow-up.
Time Frame: Week 0, week 40
Population: The FAS included all randomized participants. Number analyzed=number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 481 | 480
Kilogram (kg)
  On-treatment without rescue medication: number analyzed (Participants) | 425 | 434
  On-treatment without rescue medication | -6.0 (5.8) | -7.0 (5.8)
  In-trial: number analyzed (Participants) | 467 | 457
  In-trial | -5.7 (5.9) | -6.7 (5.9)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) to week 40 in FPG was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first.
Time Frame: Week 0, week 40
Population: The FAS included all randomized participants. Overall number of participants analyzed=number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 423 | 429
Millimoles per liter (mmol/L) | -3.2 (2.8) | -3.4 (3.1)

4. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change from baseline (week 0) to week 40 in BMI was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first.
Time Frame: Week 0, week 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram per squaremeter (Kg/m^2)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 425 | 434
Kilogram per squaremeter (Kg/m^2) | -2.1 (2.1) | -2.5 (2.1)

5. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) to week 40 in waist circumference was evaluated. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first.
Time Frame: Week 0, week 40
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 423 | 433
Centimeter (cm) | -5.2 (6.1) | -5.9 (6.2)

6. Secondary Outcome: Participants Who Achieved HbA1c < 7.0%
Description: Percentage of participants who achieved HbA1c < 7.0% is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first. Missing HbA1c assessment at week 40 was imputed using observed data from participants within same treatment group.
Time Frame: Week 40
Population: The FAS included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 481 | 480
Percentage of participants | 57.5 | 67.6

7. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5%
Description: Percentage of participants who achieved HbA1c ≤ 6.5% is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first. Missing HbA1c assessment at week 40 was imputed using observed data from participants within same treatment group.
Time Frame: Week 40
Population: The FAS included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 481 | 480
Percentage of participants | 38.5 | 51.7

8. Secondary Outcome: Participants Who Achieved Weight Loss ≥5%
Description: Percentage of participants who achieved weight loss ≥5% is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first. Missing body weight assessment at week 40 was imputed using observed data from participants within same treatment group.
Time Frame: Week 40
Population: The FAS included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 481 | 480
Percentage of participants | 51.3 | 59.2

9. Secondary Outcome: Participants Who Achieved Weight Loss ≥10%
Description: Percentage of participants who achieved weight loss ≥10% is presented. Results are based on the 'on-treatment without rescue medication' observation period, which started at the date of first dose of trial product to either first initiation of rescue medication or the day of last dose of trial product, whichever came first. Missing body weight assessment at week 40 was imputed using observed data from participants within same treatment group.
Time Frame: Week 40
Population: The FAS included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 481 | 480
Percentage of participants | 22.6 | 28.4

10. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Hypoglycaemic episodes defined as treatment-emergent if the onset of the episode occurs within the on-treatment observation period. Severe or BG-confirmed symptomatic hypoglycaemia is an episode that required assistance from another person for recovery and blood glucose-confirmed by a plasma glucose value <3.1 mmol/L (56 milligrams per deciliter (mg/dL)) with symptoms consistent with hypoglycaemia. Results are based on the 'on-treatment' observation period, which started at the date of first dose of trial product and ended at the first date of any of the following: the follow-up visit (week 47), the treatment discontinuation follow-up visit (end of treatment + 7 weeks), the date of last dose of trial product +49 days or the end-date for the 'in-trial' observation period.
Time Frame: Week 0 to week 47
Population: The SAS included all participants exposed to at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 480 | 479
Episodes | 28 | 21

11. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) to week 40 in pulse rate is presented. Results are based on the 'on-treatment' observation period, which started at the date of first dose of trial product and ended at the endpoint-specific end-date.
Time Frame: Week 0, week 40
Population: The SAS included all participants exposed to at least one dose of trial product. Overall number of participants analyzed=number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
Number analyzed (Participants) | 444 | 442
Beats per minute | 2.8 (10.0) | 3.3 (9.5)

ADVERSE EVENTS:
Time Frame: Weeks 0-47
Description: All presented AEs are TEAEs. A TEAE was defined as an event that had onset during the on-treatment period. Results are based on the SAS which comprised of all participants exposed to at least one dose of trial product.
Arm/Group | Semaglutide 1.0 mg | Semaglutide 2.0 mg
All-Cause Mortality (participants affected / at risk) | 1/480 | 2/479
Serious Adverse Events (participants affected / at risk) | 25/480 | 21/479
Other Adverse Events (participants affected / at risk) | 126/480 | 132/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=480) | Semaglutide 2.0 mg (N=479)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 3 (3) | 0 (0)
Death; reason unknown (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Smear cervix abnormal (Investigations) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=480) | Semaglutide 2.0 mg (N=479)
Decreased appetite (Metabolism and nutrition disorders) | 18 (18) | 29 (29)
Diarrhoea (Gastrointestinal disorders) | 42 (83) | 45 (51)
Dyspepsia (Gastrointestinal disorders) | 25 (26) | 16 (17)
Nausea (Gastrointestinal disorders) | 70 (98) | 69 (98)
Vomiting (Gastrointestinal disorders) | 32 (40) | 37 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT03989232/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03989232/SAP_002.pdf